CLINICAL TRIAL: NCT06498037
Title: Optimizing Subcutaneous FEntanyl titRation: RApid Achievement of Adequate Exposure When Treating Cancer-Related paIn.
Acronym: FERRARI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Prof. R.H.J. Mathijssen, MD, PhD, prof.R.H.J. Mathijssen, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-507355-30
Record Dates: First submitted 2024-06-26; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Cancer Pain
MeSH Terms: conditions — Cancer Pain | interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: a single-arm PK-study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental): Patients are given loading doses when dose-increasing fentanyl. The concentrations at 12 and 48 hours after dose increase will be compared
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Administration of subcutaneously administered fentanyl loading boluses

SUMMARY:
The primary objective is to evaluate the effect of loading boluses when dose incresaing treatment with SC fentanyl in patients with cancer. The primary endpoint of this study is to prove the non-inferiority of fentanyl plasma concentrations 12 hours after dose augmentation compared to 48 hours after dose augmentation within each patient.

Patients will be treated with additional loading boluses and plasma-PK samples will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Able to understand the written information and able to give informed consent.
* Current or planned treatment with SC fentanyl for cancer-related pain

Exclusion Criteria:

* Pregnancy or/ and breastfeeding
* Other ways of using fentanyl (sublingual, nasal spray and oromucosal)
* Liver function CPS B or C
* The use of strong CYP3A4 inhibitors of inducers [9]
* Presence of somnolence, respiratory depression or CTCAE grade 2 adverse events.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint of this study is to prove the non-inferiority in fentanyl plasma concentrations 12 hours after dose augmentation compared to 48 hours after dose augmentation within each patient using a bioequivalence approach | 48 hours after dose increase
  Using a paired t-test the geometric mean of the ratio of the two fentanyl plasma concentrations will be compared. The 90% confidence interval of the geomteric mean should fall within the range of 80 - 125%.

SECONDARY OUTCOMES:
Investigate the safety of the loading bolus strategy by assessing whether CTCAE grade III or higher occur as a consequence of the fentanyl loading boluses. | up to 48 hours after dose increase
  This will be performed as a descriptive analysis
Describe the course of patient reported pain intensity in the 48 hours following the loading boluses. | up to 48 hours after dose increase
  This will be performed as a descriptive analysis
Accurately assess the rate of fentanyl absorption after SC fentanyl administered as a bolus. | up to 48 hours after dose increase
  The pharmacokinetic data will be imputed into a population pharmacokinetic model that allows to simulate other situations and dosing regimens which will be used to further optimize dosing of subcutaneously administered fentanyl

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No